CLINICAL TRIAL: NCT03397277
Title: Preparing for the Worst - Promoting Safety Behaviours in Antenatal Care Among Norwegian, Pakistani and Somali Pregnant Women
Brief Title: Promoting Safety Behaviours in Antenatal Care Using a Video
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo Metropolitan University (Other)
Collaborators: University of Oslo (Other); Norwegian University of Science and Technology (Other); La Trobe University (Other)
Responsible Party: Principal Investigator, Mirjam Lukasse, Professor, Oslo Metropolitan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 260355
Record Dates: First submitted 2017-10-24; First posted 2018-01-11 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Intimate Partner Violence
Keywords: IPV

STUDY DESIGN:
Intervention Model Description: Pregnant women will be screened for IPV using a modified version of the Abuse Assessment Screening. Women who screen positive are randomized into either the intervention video or a control video. Women screening negative for violence will be shown the control video. All women receive standard care and a card with high quality websites about safe pregnancy. Hidden among these is a webside that informs women about IPV (rights, safety etc..). Three months after birth all the women screening positive for violence will receive another questionnaire to fill out. In addition will a random sample of women who screened negative for IPV be asked to fill out a questionnaire at the same time. This group will be double the size of the women screening positive.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: All women will be shown a video (also women not screening positive for IPV). Unless staff ask women about the content of the video or the women discloses this, care providers will not know which film participants have viewed. As we include a group of women who screened negative for IPV in the assessment three months after birth care providers will not know who who screened positive and who screened negative. In the file the variable for control og intervention video will be blinded. Women will be selected for the post-partum questionnaire based on the screening for abuse. All abused women and for each abused woman two without abuse will be selected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Screened positive intervention video (Experimental): Safety behaviour promoting video
  Interventions: Behavioral: Safety behaviour promoting video
- Screened positive control video (Sham Comparator): Pregnant women who screen positive for IPV using the AAS who are randomized into viewing the control video
  Interventions: Behavioral: Control video

INTERVENTIONS:
Behavioral: Safety behaviour promoting video — A 7 min. video which teaches 15 different safety behaviours to reduce violence or the effect of violence
  Arms: Screened positive intervention video
Behavioral: Control video — A 7 min. video which teaches women about safety regarding food, alcohol, smoking, medication and physical activity during pregnancy
  Arms: Screened positive control video

SUMMARY:
This study investigates the effect of a video which teaches 15 safety behaviours for women subject to intimate partner violence (IPV) during pregnancy. Half of the women screening positive for IPV during pregnancy will view the intervention video. The other half will view a control video.

DETAILED DESCRIPTION:
Intimate partner violence (IPV) poses a risk for the health of the woman during pregnancy also for the health of the unborn child. Pregnancy is time when nearly all women have regular contact with the healthcare system. Pregnancy is also a time during which women consider their situation and are open for change.

Healthcare staff have the opportunity to ask pregnant women if they experience IPV and need to know how to respond to women experiencing IPV. Healthcare staff can refer to other services. If staff are uncertain if referral is needed or wanted they can teach women how to increase their own safety and prepare for leaving through a number of safety promoting behaviours.The safety behaviours were originally developed in the USA to counsel women who attended a family violence unit and qualified for a protection order.

Women do not always disclose the true nature of their IPV to staff. However, they could still benefit from learning about safety promoting behaviours. Using a video for teaching allows for the use of pictures and sound and options for several languages.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women attending antenatal care at the community health center,
* 18 years or older,
* understanding sufficient Norwegian, Urdu, Somali or English to complete the questionnaire and understand the video.

Exclusion Criteria:

* women who do not speak or understand the languages provided in the study (English, Urdu, Somali and Norwegian)
* women who have never been in an adult intimate relationship
* women who are closely attended by male partner
* women who do not have the mental of physical capacity to answer the questionnaire.
* women who cannot fill out the questionnaire in privacy

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only women are pregnant so only women can be recruited to this study
Enrollment: 250 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
Adoption of safety behaviours | change from pregnancy to 3 months postpartum
  Number of used safety behaviours
The World Health Organisation Quality of Life Brief (WHOQOL-BREF) | Change from pregnancy to 3 months postpartum
  A scale of 26 items assessing four dimensions of quality of life (QOL), physical, psychological, environmental and social. Low score equals low QOL. Mean scores are calculated for each domain.

SECONDARY OUTCOMES:
Prevalence of Intimate Partner Violence (IPV) measured using Composite Abuse Scale (revised) - Short Form (CAS R SF) | change from pregnancy to 3 months postpartum
  CAS(R)-SF is a 15-item instrument capturing physical, sexual and psychological abuse and overall IPV. Total score ranges from 0 to 75. Low score indicates less violence. Mean total score is calculated and compared.
Symptoms of depression | Change from pregnancy to 3 months postpartum. Minimum score is 0, maximum score is 15. The lower the score the fewer symptoms of depression the person has. A cut-off of 7 or more is used to indicate symptoms of depression.
  Edinburgh Depression Scale -5 (short version)

OTHER OUTCOMES:
Mode of delivery | at birth
  operative delivery vs. spontaneous vaginal birth
Birth weight | at birth
  neonates birthweight in grams
Initiation and early cessation of breastfeeding | approximately 3 months postpartum
  We will use 3 questions developed for the Norwegian Mother and Child Cohort Study (MoBa) which recruited approx 100.000 women. These questions have been developed by nutrionalists and have been used in studies and published in relation to abuse, BMJ Open. 2015 Dec 18;5(12):e009240. doi: 10.1136/bmjopen-2015-009240. Past and recent abuse is associated with early cessation of breast feeding: results from a large prospective cohort in Norway.The questions allows for measuring the proportion of women initiating breastfeeding and how many stopped breastfeeding by the time of measurement postpartum
Method of pain relief used during labour | at birth
  we will record the number of women in each arm who receive epidural analgesia, pudendal analgesia, used water immersion for pain relief, used nitrous oxide inhalation, used other methods.
birth experience | 3 months postpartum
  One question asking if the birth experience was solely positive, positive with negative elements, negative with positive elements or solely negative. This question has been used in other studies and the answering options are usually dichotomised into a positive or negative birth experience

CONTACTS AND LOCATIONS:
Overall Officials: Mirjam Lukasse, PhD, Principal Investigator — Oslo and Akershus University College
Locations (19):
- Norway (19):
  - Trøgstad Community Health Center, Askim
  - Nordberg, Ås
  - Ås Community Health Center, Ås
  - Rælingen Community Health Center, Flateby
  - Familie Hus Halden, Halden
  - Aurskog- Høland Community Health Center, Høland
  - Jevnaker Community Health Center, Jevnaker
  - Lillestrøm Communicy Health Center, Lillestrøm
  - Nesodden Community Health Center, Nesoddtangen
  - Oppegård Community Health Center, Oppegård
  - Grorud Community Health Center, Oslo
  - Bjerke Community Center, Oslo
  - Health Centre Alna, Oslo
  - Stovner Community Health Center, Oslo
  - Rakkestad Community Health Center, Rakkestad
  - Skedsmo Community Health Center, Skedsmokorset
  - Langhus, Ski
  - Ski Community Health Center, Ski
  - Våler Community Health Center, Våler

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Flaathen EME, Henriksen L, Smastuen MC, Schei B, Taft A, Noll J, Garnweidner-Holme L, Lukasse M. Safe Pregnancy intervention for intimate partner violence: a randomised controlled trial in Norway among culturally diverse pregnant women. BMC Pregnancy Childbirth. 2022 Feb 21;22(1):144. doi: 10.1186/s12884-022-04400-z. PMID 35189843
- [Derived] Walter B, Indreboe H, Lukasse M, Henriksen L, Garnweidner-Holme L. Pregnant Women's Attitudes Toward and Experiences With a Tablet Intervention to Promote Safety Behaviors in a Randomized Controlled Trial: Qualitative Study. JMIR Form Res. 2021 Jul 20;5(7):e28680. doi: 10.2196/28680. PMID 34283023
- [Derived] Garnweidner-Holme L, Henriksen L, Flaathen EM, Klette Bohler T, Lukasse M. Midwives' Attitudes Toward and Experience With a Tablet Intervention to Promote Safety Behaviors for Pregnant Women Reporting Intimate Partner Violence: Qualitative Study. JMIR Mhealth Uhealth. 2020 May 20;8(5):e16828. doi: 10.2196/16828. PMID 32432553
- [Derived] Henriksen L, Flaathen EM, Angelshaug J, Garnweidner-Holme L, Smastuen MC, Noll J, Taft A, Schei B, Lukasse M. The Safe Pregnancy study - promoting safety behaviours in antenatal care among Norwegian, Pakistani and Somali pregnant women: a study protocol for a randomized controlled trial. BMC Public Health. 2019 Jun 10;19(1):724. doi: 10.1186/s12889-019-6922-y. PMID 31182062

DOCUMENTS (3):
  • Study Protocol (2017-12-29): https://cdn.clinicaltrials.gov/large-docs/77/NCT03397277/Prot_001.pdf
  • Statistical Analysis Plan (2017-12-29): https://cdn.clinicaltrials.gov/large-docs/77/NCT03397277/SAP_002.pdf
  • Informed Consent Form (2018-01-11): https://cdn.clinicaltrials.gov/large-docs/77/NCT03397277/ICF_003.pdf